CLINICAL TRIAL: NCT03635242
Title: Characterization by Clinimetric Indicators of Chronic Low Back Pain Subjects Versus Post-treatment Healed Patients by Therapeutic Exercise
Brief Title: Characterization by Clinimetric Indicators of Chronic Low Back Pain Subjects Versus Healed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Alejandro Caña Pino, Medical Surgical-Therapy Department, Universidad de Extremadura Facultad de Medicina, Badajoz, Spain, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08062018
Record Dates: First submitted 2018-08-10; First posted 2018-08-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Chronic Low Back Pain; Postural Low Back Pain
Keywords: postural control; Chronic Low Back Pain; therapeutic excercise; healed patients
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control. no therapeutic program (Active Comparator): The control group continued to perform their daily activities without changing any habit. Group of healthy subjects Assessment of postural control through accelerometry and pressure platform
  Interventions: Other: Control. no therapeutic program
- Experimental. Therapeutic program (Experimental): People with chronic back pain of at least 3 months duration, to whom the therapeutic exercise of motor control and pain education based on neuroscience will be applied 2 days a week for 2 months.
  Prior to the intervention, a postural control assessment will be made by accelerometry and pressure platform
  Interventions: Other: Experimental. Therapeutic program

INTERVENTIONS:
Other: Control. no therapeutic program — The control group continued to perform their daily activities without changing any habit. Group of healthy subjects Assessment of postural control through accelerometry and pressure platform
  Arms: Control. no therapeutic program
Other: Experimental. Therapeutic program — People with chronic back pain of at least 3 months duration, to whom the therapeutic exercise of motor control and pain education based on neuroscience will be applied 2 days a week for 2 months.
  Prior to the intervention, a postural control assessment will be made by accelerometry and pressure platform
  Arms: Experimental. Therapeutic program

SUMMARY:
Pretending with the use of accelerometers and pressure platform, determine indicators that are useful to therapists to assess postural control and balance, to subsequently allow to evaluate the effect of therapeutic interventions through therapeutic exercise of motor control in patients with chronic low back pain .

DETAILED DESCRIPTION:
The records are made simultaneously with the different evaluation equipment, accelerometer and pressure platform. The tests are performed in a control group of healthy subjects, and in an experimental group with DLC receiving a program of therapeutic exercise based and pain education based on neuroscience.

After the collection of the records, the behavior patterns in both groups are evaluated, the possible differences among them are established for the clinimetric indicators analyzed related to the postural control, as well as a characteristic of the sample.

Subsequently, through the evaluation after the intervention of the experimental group we will analyze the effect of a physiotherapy treatment based on the therapeutic exercise of motor control on parameters related to postural control and clinical variables (perceived pain, mechanosensitivity, disability and proprioceptive repositioning of the lumbar spine )

ELIGIBILITY:
Inclusion Criteria:

* low back pain with painful perception on a daily or almost daily basis for more than three months of clinical course, with or without pain radiating to the lower extremities above the knee.
* not having metal implants in the spine
* own ability to read and write
* and access the study voluntarily.

Exclusion Criteria:

* vestibular disorders
* without severe visual impairment
* no medication intake with a potential effect on balance during the 90 days prior to data collection
* physiotherapy treatment 2 weeks before the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
pressure platform and accelerometry | 4 weeks
  Stay for 30 seconds each test on a pressure platform. Accelerometer in the pelvis (center of mass), fixed by velcro tape. Application of the Romberg test. (Standing with open eyes and closed on stable and unstable surface).The unit of the accelerometer is mg (1 mg = 0.001) and the kinetic energy of the signal is measured in Julians x 10-6 The displacement unit of the pressure center of the platform is millimeters

SECONDARY OUTCOMES:
weight | 4 weeks
  Descriptive variable. Its unit of measurement is Kilograms
Height | 4 weeks
  Descriptive variable. Its unit of measurement is meters
age | 4 weeks
  Descriptive variable. Its unit of measurement is years
EVA (Visual Analog Scale). | 4 weeks
  Used for pain assessment in an analogical way, that is, by means of a line of 10 centimeters. 0 (absence of pain); 10 (maximum pain)
Algometry | 4 weeks
  Algometry at 5 cm from the spinous process of L3 and in lateral epicondyl (Bilateral)
Joint Position Sense (JPS) | 4 weeks
  Joint Position Sense (JPS) to evaluate the proprioceptive joint positioning of the lumbar spine with a digital goniometer at 30º flexion in standing and sitting
Roland Morris | 4 weeks
  determine the degree of disability. The extreme values oscillate between 0 (absence of disability due to low back pain) and 24 (maximum possible disability)
Oswestry Disability Index | 4 weeks
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability
  Scoring instructions For each section of the total possible score is 5: if the first statement is mark ed the section score = 0; if the last statement is marked, it = 5.
Pain Catastrophizing Scale (PCS) | 4 weeks
  it measures the catastrophic thoughts before the pain, that is, the negative thought before the pain. In the PCS, people take the painful past experience as a reference and indicate the degree to which they experience certain thoughts and feelings. The PCS is composed of 13 items, on a Likert scale of 5 points that goes from 0 (never) to 4 (always).
  Higher scores indicate higher levels of catastrophism
The Tampa Kinesiofobia Scale (TSK) | 4 weeks
  It is commonly used in clinical practice to quantify pain levels related to fear of activity or to a new injury in patients with back pain. Patients with high levels of kinesiofobia are often considered at greater risk of developing long-term activity limitation and chronicity

CONTACTS AND LOCATIONS:
Overall Officials: Luis LE Espejo-Antúnez, PhD, Study Director — Universidad de Extremadura. Facultad de Medicina (Badajoz). Spain; Mª Dolores MD Apolo-Arenas, PhD, Study Director — Universidad de Extremadura. Facultad de Medicina (Badajoz). Spain; Alejandro Caña-Pino, PT,MSc, Principal Investigator — Universidad de Extremadura. Facultad de Medicina (Badajoz). Spain
Locations (1):
- Universidad de Extremadura, Badajoz, Spain